CLINICAL TRIAL: NCT05791994
Title: Effet d'Exercices Visuels de Stimulation Cognitive Sur Les capacités Attentionnelles Chez la Personne âgée (Etude Pilote)
Brief Title: EVASION: Effect of VisuAl Stimulation on attentION
Acronym: EVASION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-A00235-40
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Geriatrics; Cognitive impairment; Visual stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Procedure: Visual cognitive stimulation exercises
- Comparator group (Active Comparator)
  Interventions: Procedure: Broadcast of a television program

INTERVENTIONS:
Procedure: Visual cognitive stimulation exercises — Patients included in Intervention group will receive a 30-minute session of complex visual stimuli on a touch screen (3 10-minute exercises : saccade exercises, then pursuit exercises, then matching exercises) every other day for 30 days, with increasing difficulty of the exercises as the sessions progress.
  Arms: Intervention group
Procedure: Broadcast of a television program — Patients included in Comparator group will watch a 30-minute television program (Allô Docteurs) on a touch screen every other day for 30 days.
  Arms: Comparator group

SUMMARY:
The main objective is to compare changes in information processing speed after 30 days of intervention in participants with a dysexecutive mild cognitive impairment (MCI) and receiving either cognitive stimulation by adapted visual exercises (Emeraude® software) or the broadcasting of a television program without cognitive stimulation.

Secondary objectives are:

* To compare, after 30 days of intervention, in participants with a dysexecutive MCI and receiving either cognitive stimulation by adapted visual exercises (Emeraude® software), or the broadcasting of a television program without cognitive stimulation :
* changes in information processing speed of each subtest,
* changes in cognitive performance,
* changes in executive functions,
* changes in walking performance.
* To compare the quality of life, after 30 days of intervention, of participants with a dysexecutive MCI and receiving either cognitive stimulation by adapted visual exercises (Emeraude® software) or the broadcasting of a television program without cognitive stimulation.
* In the "Intervention" group, to study correlations between changes in information processing speed index and the final level reached for each cognitive stimulation exercise.

DETAILED DESCRIPTION:
Attentional abilities are among the cognitive functions that are most frequently and earliest altered during aging, particularly in the case of neurodegenerative diseases such as Alzheimer's disease. This decline can be the cause of a cognitive complaint in the patient or his relatives from the prodromal stage of the disease. This mild cognitive impairment is not sufficiently advanced to have an impact on independence and autonomy, even though recent studies have reported an early modification of walking in this population, in particular in the case of a dysexecutive MCI. The current challenge is to develop strategies to prevent cognitive decline in these patients with MCI and to avoid conversion to major neurocognitive disorders. However, while "memory workshops" are offered to patients with amnestic MCI, no strategy is clearly identified for dysexecutive MCI.

Interestingly, the integration of sensory information is modified in patients with neurodegenerative diseases, and in particular visuomotor difficulties in the early stages. Measurements of evoked potentials during visual stimulation have shown that sensory responses are preserved but cognitive responses are reduced in patients with MCI. Based on this observation, an American team recently tested the effectiveness of computer-assisted visual cognitive exercises performed regularly for 8 weeks in patients without dementia, and reported an improvement in information processing speed and walking performance. These results lead us to hypothesize that regular cognitive stimulation exercises using adapted visual exercises could improve the attentional capacities and in particular the information processing speed (=mental speed) of elderly people with a dysexecutive MCI.

A complex brain stimulation software Emeraude® has recently been developed by the Centre Régional Basse Vision in Angers from a software used for more than 30 years in people with visual impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Diagnosis of mild cognitive impairment of a dysexecutive or multidomain dysexecutive nature, according to Winblad consensus criteria
* Presence of an informal caregiver
* Subject gave and signed informed consent to participate in the study
* Affiliation to a social security scheme

Exclusion Criteria:

* Presence of severe depressive symptoms (4-item Geriatric Depression Scale score > 2)
* Ophthalmological or central pathology that may affect the performance of stimulation exercises
* Regular use of psychotropic drugs that may have an impact on the performance of stimulation exercises, in the opinion of the investigator (benzodiazepines, antidepressants, neuroleptics, hypnotics)
* Use of anticonvulsant drugs
* Existence of a confusional syndrome
* Participation in another simultaneous clinical trial
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person subject to a legal protection measure
* Person unable to give consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in information processing speed | Baseline and after 30 days of intervention
  Changes in information processing speed is assessed by processing speed index

SECONDARY OUTCOMES:
Changes in information processing speed of each subtest | Baseline and after 30 days of intervention
  This outcome is assessed by Symbol Search end Coding scores
Changes in cognitive performance | Baseline and after 30 days of intervention
  This outcome is assessed by ADAS-cog score
Changes in executive functions (cognitive flexibility) | Baseline and after 30 days of intervention
  Cognitive flexibility is measured by time needed to perform the Trail-Making Test (TMT) part B minus A
Changes in executive functions (cognitive inhibition) | Baseline and after 30 days of intervention
  Cognitive inhibition is measured by time needed to perform the interference task minus the time needed to perform the denomination task
Changes in executive functions (working memory updating) | Baseline and after 30 days of intervention
  Working memory updating is assessed by digit span test
Changes in walking performance | Baseline and after 30 days of intervention
  Changes in walking performance is assessed by changes in coefficient of variation of stride time
Changes in quality of life | Baseline and after 30 days of intervention
  Quality of life is assessed by 36-Item Short Form Health Survey (SF-36)
Correlations between changes in information processing speed index and the final level reached for each cognitive stimulation exercise | After 30 days of intervention
  This outcome is assessed by the final level achieved for each cognitive stimulation exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).